CLINICAL TRIAL: NCT00224536
Title: Bone Marrow Transfer to Enhance ST-Elevation Infarct Regeneration-1
Brief Title: Bone Marrow Transfer to Enhance ST-Elevation Infarct Regeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOOST-1
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2005-09-23 (Estimated); Status verified 2005-09

CONDITIONS: Coronary Artery Disease
Keywords: Myocardial infarction; Bone marrow cells; Intracoronary
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

INTERVENTIONS:
Procedure: Intracoronary bone marrow cell transfer

SUMMARY:
After successful percutaneous coronary intervention (PCI) for acute ST-segment elevation myocardial infarction, 60 patients were randomly assigned to either a control group (n=30) that received optimum postinfarction medical treatment, or a bone-marrow-cell group (n=30) that received optimum medical treatment and intracoronary transfer of autologous bone-marrow cells 4·8 days (SD 1·3) after PCI. Primary endpoint was global left-ventricular ejection fraction (LVEF) change from baseline to 6 months' follow-up, as determined by cardiac MRI. Image analyses were done by two investigators blinded for treatment assignment. Analysis was per protocol.

Global LVEF at baseline (determined 3·5 days [SD 1·5] after PCI) was 51·3 (9·3%) in controls and 50·0 (10·0%) in the bone-marrow cell group (p=0·59). After 6 months, mean global LVEF had increased by 0·7 percentage points in the control group and 6·7 percentage points in the bone-marrow-cell group (P=0·0026).

Transfer of bone-marrow cells enhanced left-ventricular systolic function primarily in myocardial segments adjacent to the infarcted area. Cell transfer did not increase the risk of adverse clinical events, in-stent restenosis, or proarrhythmic effects.

DETAILED DESCRIPTION:
Emerging evidence suggests that stem cells and progenitor cells derived from bone marrow can be used to improve cardiac function in patients after acute myocardial infarction. In this randomised trial, we aimed to assess whether intracoronary transfer of autologous bone-marrow cells could improve global left-ventricular ejection fraction (LVEF) at 6 months' follow-up.

After successful percutaneous coronary intervention (PCI) for acute ST-segment elevation myocardial infarction, 60 patients were randomly assigned to either a control group (n=30) that received optimum postinfarction medical treatment, or a bone-marrow-cell group (n=30) that received optimum medical treatment and intracoronary transfer of autologous bone-marrow cells 4·8 days (SD 1·3) after PCI. Primary endpoint was global left-ventricular ejection fraction (LVEF) change from baseline to 6 months' follow-up, as determined by cardiac MRI. Image analyses were done by two investigators blinded for treatment assignment. Analysis was per protocol.

Global LVEF at baseline (determined 3·5 days [SD 1·5] after PCI) was 51·3 (9·3%) in controls and 50·0 (10·0%) in the bone-marrow cell group (p=0·59). After 6 months, mean global LVEF had increased by 0·7 percentage points in the control group and 6·7 percentage points in the bone-marrow-cell group (P=0·0026).

Transfer of bone-marrow cells enhanced left-ventricular systolic function primarily in myocardial segments adjacent to the infarcted area. Cell transfer did not increase the risk of adverse clinical events, in-stent restenosis, or proarrhythmic effects. Intracoronary transfer of autologous bone-marrow-cells promotes improvement of left-ventricular systolic function in patients after acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they were admitted within 5 days of the onset of symptoms of a first ST-segment elevation myocardial infarction
* Had undergone successful PCI with stent implantation in the infarctrelated artery
* Had hypokinesia or akinesia involving more than two thirds of the left-ventricular anteroseptal, lateral, and/or inferior wall, as shown by angiography done immediately after PCI.

Exclusion Criteria:

* We excluded patients who had multivessel coronary artery disease, pulmonary edema, cardiogenic shock, advanced renal or hepatic dysfunction, or documented terminal illness or cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-01; Study Completion 2003-10

PRIMARY OUTCOMES:
Left ventricular ejection fraction change between groups at month 6

SECONDARY OUTCOMES:
Safety
Left ventricular volumes
Infarct size
Subgroup analyses

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Drexler, MD, Principal Investigator — Hannover Medical School, Germany
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Result] Wollert KC, Meyer GP, Lotz J, Ringes-Lichtenberg S, Lippolt P, Breidenbach C, Fichtner S, Korte T, Hornig B, Messinger D, Arseniev L, Hertenstein B, Ganser A, Drexler H. Intracoronary autologous bone-marrow cell transfer after myocardial infarction: the BOOST randomised controlled clinical trial. Lancet. 2004 Jul 10-16;364(9429):141-8. doi: 10.1016/S0140-6736(04)16626-9. PMID 15246726